CLINICAL TRIAL: NCT00159276
Title: GR Defect in Sputum Cells in COPD
Status: Withdrawn | Type: Observational
Sponsor: Imperial College London (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D5899N00007A
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

INTERVENTIONS:
Procedure: Induced Sputum

SUMMARY:
To investigate a possible mechanism of the GR defect in patients with severe COPD by studying the effect of dexamethasone (Dex) on GR-GRE binding, expression of inflammatory and anti-inflammatory factors such as IL-6, IL-8, MKP-1, GILZ, SLPI production in sputum cells

ELIGIBILITY:
Inclusion Criteria:

* Patients with moderate (stage II, GOLD) COPD or subjects who are healthy smokers or subjects who are non-smokers.
* Written informed consent

Exclusion Criteria:

* Current upper respiratory tract infections
* Any significant disease or disorder (e.g. cardiovascular, pulmonary (other than asthma), gastrointestinal, liver, renal, neurological, musculoskeletal, endocrine, metabolic, malignant, psychiatric, major physical impairment) which, in the opinion of the investigator, may either put the subject at risk because of participation in the study, or may influence the results of the study, or the subjects ability to participate in the study
* Subjects not considered capable, as judged by the investigator, of following instructions of the study, e.g. because of a history of alcohol or drug abuse or any other reason

Ages: 35 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2005-12 (Estimated); Primary Completion 2005-12 (Estimated); Study Completion 2005-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Sergei A Kharitonov, MD PhD, Principal Investigator — Imperial College London
Locations (1):
- Section of Airway Disease, Asthma Lab, Imperial College London, Royal Brompton Hospital, London, United Kingdom